CLINICAL TRIAL: NCT06706843
Title: The Effect of Transtheoretical Model-based Motivational Interview on Self-efficacy and Illness Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HÜSEYİN ÇAPUK (Other)
Responsible Party: Sponsor-Investigator, HÜSEYİN ÇAPUK, Assoc. Prof., Şırnak Üniversitesi
Organization: Şırnak Üniversitesi (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 112
Record Dates: First submitted 2024-09-27; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hemodialysis Units, Hospital

STUDY DESIGN:
Intervention Model Description: Transtheoretical Model Based Motivational interview was conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- motivational interview group (Experimental): This group received motivational interviewing training based on the transtheoretical model.
  Interventions: Behavioral: Transtheoretical Model Based Motivational Interviewing; Other: routine clinical care
- control group (Experimental): No intervention was performed. Patients continued their routine treatment.
  Interventions: Other: routine clinical care

INTERVENTIONS:
Behavioral: Transtheoretical Model Based Motivational Interviewing — Transtheoretical Model Based Motivational Interviewing was applied to haemodialysis patients in 6 sessions.
  Arms: motivational interview group
Other: routine clinical care — routine clinical care

SUMMARY:
Aim: This study was planned to determine the effect of transtheoretical model-based motivational interviewing on patients' self-efficacy and disease adherence in patients receiving haemodialysis treatment.

Study design and methods: This study was conducted between June 2022 and April 2023 according to the experimental research model with pre-test and post-test control group. The research was completed with a total of 60 hemodialysis patients, 30 in the experimental group and 30 in the control group.

ELIGIBILITY:
Inclusion Criteria:

Being on hemodialysis treatment Being able to read and writeH

Exclusion Criteria:

Not knowing how to read or write, Having a psychological disorder that prevents speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Results | Time Frame: six weeks
  A transtheoretical model-based motivational interview was applied to hemodialysis patients in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Rukuye Aylaz, Prof. Dr., Study Director — İnönü Üniversitesi
Locations (1):
- Inonu University, Malatya, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Capuk H, Aylaz R. The Impact of Transtheoretical Model-Based Motivational Interviewing on Self-Efficacy and Adherence to Treatment in Hemodialysis Patients. J Eval Clin Pract. 2025 Jun;31(4):e70152. doi: 10.1111/jep.70152. PMID 40492930